CLINICAL TRIAL: NCT01690663
Title: Dose Response Study of Dexamethasone in Combination With Bupivacaine 0.25% in Ultrasound Guided Supraclavicular Brachial Plexus Nerve Block, a Randomized, Placebo Controlled Prospective Clinical Trial
Brief Title: Dose Response Study of Dexamethasone in Combination With Bupivacaine 0.25%
Acronym: Dex Dose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 815628
Record Dates: First submitted 2012-09-12; First posted 2012-09-24 (Estimated); Results first posted 2017-05-04 (Actual); Last update posted 2017-05-04 (Actual); Status verified 2017-03

CONDITIONS: Post Surgical Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Dexamethasone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Bupivacaine 0.25% mixed with 1ml normal saline (Placebo Comparator): Bupivacaine 0.25% mixed with 1ml normal saline (placebo/control group)
  Interventions: Drug: Bupivacaine 0.25%; Drug: normal saline
- Bupivacaine 0.25% with 1mg dexamethasone (1ml) (Active Comparator): Bupivacaine 0.25% mixed with 1mg preservative free dexamethasone (1ml)
  Interventions: Drug: Bupivacaine 0.25%; Drug: Dexamethasone
- Bupivacaine 0.25% mixed with 2mg dexamethasone (Active Comparator): Bupivacaine 0.25% mixed with 2mg preservative free dexamethasone (1ml)
  Interventions: Drug: Bupivacaine 0.25%; Drug: Dexamethasone
- Bupivacaine 0.25% mixed with 4mg dexamethasone (1ml (Active Comparator): Bupivacaine 0.25% mixed with 4mg preservative free dexamethasone (1ml
  Interventions: Drug: Bupivacaine 0.25%; Drug: Dexamethasone

INTERVENTIONS:
Drug: Bupivacaine 0.25%
Drug: Dexamethasone
  Arms: Bupivacaine 0.25% mixed with 2mg dexamethasone; Bupivacaine 0.25% mixed with 4mg dexamethasone (1ml; Bupivacaine 0.25% with 1mg dexamethasone (1ml)
Drug: normal saline — placebo
  Arms: Bupivacaine 0.25% mixed with 1ml normal saline

SUMMARY:
When used in conjunction with a local anesthetic, dexamethasone may prolong both the sensory and motor effects of high supraclavicular brachial plexus nerve block (SBP) in arthroscopic shoulder surgery. This study seeks to determine if there is a relationship between the duration of sensory and motor blockade in supraclavicular brachial plexus nerve blocks (SBP) when combined with increasing doses of dexamethasone.

DETAILED DESCRIPTION:
The exact mechanism of dexamethasone on peripheral nerve block is unclear. The current theory is that the effect is not dose related, while only 4mg and 8mg doses were studied. Our hypothesis is that the dose differences at 1mg, 2mg, or 4mg, does not have significant effect on the duration of analgesia. Therefore, we are not considering any patients to receive suboptimal dosing of preservative free dexamethasone in this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 70 scheduled for primary shoulder arthroscopy who have already elected to receive and are eligible for regional anesthesia (brachial plexus nerve block) prior to consenting for study.
2. Ability to sign informed consent.
3. Ability to follow study protocol, and speak, read and write in English.
4. Must have valid phone number for follow-up purpose.
5. Must be able to receive all protocol medications to include the dexamethasone, ketorolac, hydromorphone, and percocet.

Exclusion Criteria:

1. Patient younger than 18 years old and older than age 70
2. Patient refusal to sign consent
3. Chronic opioid use (defined as narcotic use longer than 3 months) as documented in patient's medical record
4. Allergy to any of the protocol medications
5. Patients with severe lung disease, contra lateral phrenic nerve injury, insulin-dependent diabetes, hepatic disease/failure, kidney disease/failure as documented in patient's medical record
6. Pregnancy (positive urine pregnancy test result in Preop area on morning of surgery)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jiabin Liu, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Presbyterian Medical Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine 0.25% Mixed With 1ml Normal Saline: Bupivacaine 0.25% mixed with 1ml normal saline (placebo/control group)
  Bupivacaine 0.25%
  normal saline: placebo
- Bupivacaine 0.25% With 1mg Dexamethasone (1ml): Bupivacaine 0.25% mixed with 1mg preservative free dexamethasone (1ml)
  Bupivacaine 0.25%
  Dexamethasone
- Bupivacaine 0.25% Mixed With 2mg Dexamethasone: Bupivacaine 0.25% mixed with 2mg preservative free dexamethasone (1ml)
  Bupivacaine 0.25%
  Dexamethasone
- Bupivacaine 0.25% Mixed With 4mg Dexamethasone (1ml: Bupivacaine 0.25% mixed with 4mg preservative free dexamethasone (1ml
  Bupivacaine 0.25%
  Dexamethasone
Period: Overall Study
Arm/Group | Bupivacaine 0.25% Mixed With 1ml Normal Saline | Bupivacaine 0.25% With 1mg Dexamethasone (1ml) | Bupivacaine 0.25% Mixed With 2mg Dexamethasone | Bupivacaine 0.25% Mixed With 4mg Dexamethasone (1ml
Started | 23 | 20 | 22 | 24
Completed | 20 | 17 | 19 | 20
Not Completed | 3 | 3 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine 0.25% Mixed With 1ml Normal Saline | Bupivacaine 0.25% With 1mg Dexamethasone (1ml) | Bupivacaine 0.25% Mixed With 2mg Dexamethasone | Bupivacaine 0.25% Mixed With 4mg Dexamethasone (1ml | Total
Number analyzed (Participants) | 23 | 20 | 22 | 24 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 23 | 20 | 22 | 24 | 89
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.1 (11.3) | 46.2 (11.8) | 48.8 (14.1) | 53.0 (12.5) | 48.4 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 6 | 5 | 22
  Male | 18 | 14 | 16 | 19 | 67
Region of Enrollment [Number; unit: participants]
  United States | 23 | 20 | 22 | 24 | 89
BMI [Mean (Standard Deviation); unit: kg/m2] | 30.4 (6.6) | 29.4 (4.0) | 28.9 (4.4) | 31.0 (6.3) | 30.3 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome Variable is Post Operative Sensory Block Duration
Description: This is defined as time from the completion of the block to the initiation of supplemental analgesia medications after hospital discharge. The patients were evaluated on different days to capture the exact end time, which was the initiation of supplemental analgesia medication. We intentionally contacted patients several times to capture the time as early as possible to minimize recall bias.
Time Frame: days 1, 2, and day 7
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | Bupivacaine 0.25% Mixed With 1ml Normal Saline | Bupivacaine 0.25% With 1mg Dexamethasone (1ml) | Bupivacaine 0.25% Mixed With 2mg Dexamethasone | Bupivacaine 0.25% Mixed With 4mg Dexamethasone (1ml
Number analyzed (Participants) | 20 | 17 | 19 | 20
hours | 12.1 [9.8 to 20.9] | 22.3 [19.0 to 24.9] | 23.3 [19.5 to 26.8] | 21.2 [16.8 to 23.9]

2. Secondary Outcome: The Secondary Outcome Variable is Post Operative Motor Block Duration
Description: This is defined as time from the completion of the block to the time when patient is able to move his or her forearm and/or hands. The patients were evaluated on different days to capture the exact end time, which was the initiation of supplemental analgesia medication. We intentionally contacted patients several times to capture the time as early as possible to minimize recall bias.
Time Frame: days 1, 2, and day 7
Measure: Mean (Inter-Quartile Range); unit: hours
Arm/Group | Bupivacaine 0.25% Mixed With 1ml Normal Saline | Bupivacaine 0.25% With 1mg Dexamethasone (1ml) | Bupivacaine 0.25% Mixed With 2mg Dexamethasone | Bupivacaine 0.25% Mixed With 4mg Dexamethasone (1ml
Number analyzed (Participants) | 20 | 17 | 19 | 20
hours | 12.1 [8.9 to 19.4] | 21 [16.8 to 22.7] | 20.9 [16.1 to 23.7] | 19.4 [14.9 to 23.2]

ADVERSE EVENTS:
Arm/Group | Bupivacaine 0.25% Mixed With 1ml Normal Saline | Bupivacaine 0.25% With 1mg Dexamethasone (1ml) | Bupivacaine 0.25% Mixed With 2mg Dexamethasone | Bupivacaine 0.25% Mixed With 4mg Dexamethasone (1ml
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/20 | 0/22 | 0/24
Other Adverse Events (participants affected / at risk) | 0/23 | 0/20 | 0/22 | 0/24

LIMITATIONS AND CAVEATS:
First, all information was collected via telephone call during the recovery period at home, during which recall may be inaccurate. Second, we did not control the intravenous dexamethasone use, which could potentially affect the analgesia duration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes